CLINICAL TRIAL: NCT06659458
Title: Utilizing Long-read Sequencing to Investigate the EGFR Landscape of EGFR Positive Lung Cancer Patients
Acronym: EGFR Lung Canc
Status: Recruiting | Type: Observational
Sponsor: Our Lady of the Lake Hospital (Other)
Responsible Party: Principal Investigator, Leslie Son, Director of Clinical Research, Our Lady of the Lake Hospital
Other Study IDs: LSUHSCIRB_7781
Record Dates: First submitted 2024-10-23; First posted 2024-10-26 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer - Non Small Cell; EGFR Exon 19 Deletion Mutation
Keywords: Lung cancer; EGFR gene
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms | interventions — Blood Specimen Collection; Base Sequence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EGFR Positive Lung Cancer: Subjects diagnosed with EGFR positive lung cancer
  Interventions: Other: blood draw; Other: Gene sequencing
- Healthy Subjects: Subjects who do not have a cancer diagnosis
  Interventions: Other: blood draw; Other: Gene sequencing

INTERVENTIONS:
Other: blood draw — A 10ml Blood sample will be taken and used to sequence the EGFR gene and surrounding DNA.
Other: Gene sequencing — Subjects will have their DNA sequenced within and around the EGFR gene.

SUMMARY:
EGFR gene mutations are some of the most commonly occurring mutations in non-small cell lung cancer. Investigators have developed a DNA instability model that estimates a risk score to assess the likelihood of an individual acquiring a cancer-linked mutation. The aim of this study is to collect blood from both those diagnosed with EGFR positive lung cancer and healthy individuals, evaluate their gene sequence surrounding the EGFR landscape and use the cancer positive and healthy sequences to validate the risk assessment model, which may one day be used to provide insight on susceptibility of getting EGFR positive lung cancer or potentially other cancer types.

ELIGIBILITY:
Inclusion Criteria:

* 18-100 years old
* Biologically born female
* Diagnosed with EGFR positive lung cancer (Arm 1-Cancer group)
* No cancer diagnosis (Arm 2-health control)

Exclusion Criteria:

* less than 18 years of age
* Biologically born male
* Incarcerated at the time of participation

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Biologically born females
Study Population: Female adult subjects who have EGFR positive lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Differences in DNA sequence of EGFR gene | From enrollment to end of data analysis at 6 months
  Subjects who have EGFR positive lung cancer will have their gene sequence compared to those that are EGFR negative and do not have lung cancer to look for differences in the sequence.

CONTACTS AND LOCATIONS:
Locations (1):
- Our Lady of the Lake Regional Medical Center, Baton Rouge, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The demographic variables of age, race and gender will be shared with our external collaborator at Louisiana State University, Dept of Chemical Engineering in order to draw broad conclusions about the sequencing data and to use these general categories for presentation and publication. Data will be de-identified upon sharing.
Supporting Information: Study Protocol
Time Frame: The data will be available and shared with collaborators upon completion of gene sequencing analysis of the final subject and remain available until IRB closure.
Access Criteria: Only de-identified data will be shared with collaborators for the purpose of drawing conclusions and publication. Data will be sharing through a secure FileS system which is a HIPAA compliant platform offered by LSUHSC which limits access to only those for which the data is sent and does so in a secure manner.